CLINICAL TRIAL: NCT01025648
Title: A Randomized, Double-blinded or Evaluator-blinded, Placebo and Active Controlled, Six-arm, Crossover, Single Dose, Dose-ranging Study, for Initial Evaluation of Safety and Efficacy in Asthma Patients
Brief Title: Randomized, Placebo/Active Crossover Dose-ranging Study for Safety and Efficacy in Asthma Patients.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Optimization of protocol
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: API-E004-CL-A
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Asthma
Keywords: Mild to Moderate Asthma; Dyspnea; Wheezing; Status Asthmaticus
MeSH Terms: conditions — Asthma; Dyspnea; Respiratory Sounds; Status Asthmaticus | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- T1 - E004 90 mcg/actuation (Experimental): T1 - E004 (epinephrine inhalation aerosol) 90 mcg/actuation - treatment by 2 actuations of E004 at 90 mcg/actuation
  Interventions: Drug: E004 (epinephrine inhalation aerosol), 90 mcg/actuation
- T2 - E004 125 mcg/actuation (Experimental): E004 (epinephrine inhalation aerosol), 125 mcg, 2 actuations
  Interventions: Drug: E004 (epinephrine inhalation aerosol), 125 mcg
- T3 - 160 mcg/actuation (Experimental): E004 (epinephrine inhalation aerosol), 160 mcg - E004 (epinephrine inhalation aerosol), 160 mcg/ actuation, 2 actuations
  Interventions: Drug: E004 (epinephrine inhalation aerosol), 160 mcg
- T4 - 220 mcg/actuation (Experimental): E004 (epinephrine inhalation aerosol), 220 mcg - 220 mcg/actuation, 2 actuations
  Interventions: Drug: E004 (epinephrine inhalation aerosol), 220 mcg
- A - Active control (Active Comparator): epinephrine inhalation aerosol, CFC propelled 220 mcg Epinephrine Inhalation Aerosol, CFC-MDI, 2 actuations
  Interventions: Drug: epinephrine inhalation aerosol, CFC propelled
- P, Placebo HFA (Placebo Comparator): E004 placebo single treatment with 2 inhalations
  Interventions: Drug: E004 Placebo

INTERVENTIONS:
Drug: E004 (epinephrine inhalation aerosol), 90 mcg/actuation — E004 (epinephrine inhalation aerosol), 90 mcg/actuation, 2 actuations, single dose crossover, 1 -14 day washout period
  Other Names: Primatene Mist HFA
  Arms: T1 - E004 90 mcg/actuation
Drug: E004 Placebo — E004 Placebo, 0 mcg epinephrine inhalation aerosol, 2 actuations, 1 -14 day washout period
  Arms: P, Placebo HFA
Drug: E004 (epinephrine inhalation aerosol), 125 mcg — E004 (epinephrine inhalation aerosol), 125 mcg/actuation, 2 actuations, single dose crossover, 1 - 14 day washout period
  Other Names: Primatene Mist HFA
  Arms: T2 - E004 125 mcg/actuation
Drug: E004 (epinephrine inhalation aerosol), 220 mcg — E004 (epinephrine inhalation aerosol), 220 mcg - 220 mcg/actuation, 2 actuations, single dose crossover, 1 - 14 days washout period
  Other Names: Primatene Mist HFA
  Arms: T4 - 220 mcg/actuation
Drug: epinephrine inhalation aerosol, CFC propelled — epinephrine inhalation aerosol, 220 mcg/actuation, 2 actuations, single dose crossover, 1 - 14 day washout period
  Other Names: Primatene Mist
  Arms: A - Active control
Drug: E004 (epinephrine inhalation aerosol), 160 mcg — E004 (epinephrine inhalation aerosol), 160 mcg/actuation, 2 actuations, single dose crossover, 1 - 14 days washout period
  Other Names: Primatene Mist HFA
  Arms: T3 - 160 mcg/actuation

SUMMARY:
The main objective of this study is to evaluate the efficacy and safety of the Armstrong's Epinephrine HFA-MDI (E004) formulation, in comparison to the Placebo (Placebo-HFA) and an Active Control (Epinephrine CFC-MDI), and to identify the optimum E004 dose strength(s) for the ensuing pivotal clinical trials. The study will be conducted in adult patients who have intermittent, or mild-to-moderate persistent, asthma, but are otherwise healthy.

The bronchodilatory efficacy of E004, is evaluated in terms of post-dose area under the curves (AUC) of FEV1 changes (% and volumes), from the pre-dose baseline values, in comparison to the Placebo Control and the Active Control.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy, male and female adults aged 18 to 55 years at Screening.
2. Clinical diagnosis of intermittent, or mild-to-moderate persistent, asthma for at least 6 months before Screening, and having used inhaled epinephrine or β-agonist(s) for asthma control;
3. Demonstrating a baseline forced expiratory volume in 1 second (FEV1) at 50-90 percent of predicted normal at Screening;
4. Demonstrating a 12.0 percent or greater airway reversibility in FEV1 within 30 min after inhaling 2 actuations of Epinephrine CFC-MDI (440 mcg Epinephrine base) at Screening;
5. Females of child-bearing potential must be non-pregnant, non-lactating, and practicing a clinically acceptable form of birth control;
6. Demonstration of proficiency in the use of a MDI inhaler after training;
7. Having properly consented to participate in the trial.

Exclusion Criteria:

1. A smoking history of 10 or more pack-years, or having smoked within 6 months prior to Screening;
2. Upper respiratory tract infections within 2 wk, or lower respiratory tract infection within 4 wk, prior to Screening;
3. Asthma exacerbations that required emergency care or hospitalized treatment, within 4 wk prior to Screening;
4. Any current or recent respiratory conditions that, per investigator discretion, might significantly affect pharmacodynamic response to the study drugs, including cystic fibrosis, bronchiectasis, tuberculosis, emphysema, and other significant respiratory diseases besides asthma;
5. Concurrent clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine (including diabetes), psychiatric, neoplastic or other illnesses that in the opinion of the investigator could impact on the conduct, safety and evaluation of the study;
6. Known intolerance or hypersensitivity to any of the study MDI ingredients (i.e., Epinephrine, HFA-134a, CFC-12, CFC-114, polysorbate-80, ethanol, thymol, nitric acid and ascorbic acid);
7. Use of prohibited drugs or failure to observe the drug washout restrictions;
8. Having been on other investigational drug/device studies in the last 30 days prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The AUC of post-dose FEV1 percentage changes (Δ%) from the Pre-dose baseline. The primary analysis of the primary endpoint is the difference of Δ% FEV1, compared between the E004 treatment arms (T1, T2, T3 and T4) and the Placebo control (Arm P). | 360 minutes post-dose

SECONDARY OUTCOMES:
Dose response relationship of Epinephrine HFA-MDI, analyzed using efficacy data from all E004 doses. | 360 minutes post dose
AUC of FEV1 volume post-dose changes (Δ Volume) from the Pre-dose baseline. | 360 minutes post dose
Time to onset of bronchodilator effect, determined by linear interpolation as the point where FEV1 first reaches 12.0 percent from the Pre-dose Baseline. | 30 (±5) min post-dose
The peak bronchodilator response (Fmax), defined as the maximum post-dose FEV1 percent change. | 360 minutes post dose
The time to peak FEV1 effect (Tmax), defined as the time of Fmax. | 360 minutes post dose
Duration of effect, calculated as the total duration of bronchodilator effects when post-dose FEV1 reaches and stays 12.0 percent above the Pre-dose Baseline. | 360 minutes post dose
Response Rate of responders who demonstrate 12.0 percent or greater FEV1 changes from the Pre-dose baseline. | 360 minutes post dose
Vital signs, i.e., blood pressure and heart rate,at Screening baseline and 15(±5) min post dosing for reversibility | screening and 15 minutes post dose
Vital signs, i.e., blood pressure (SBP/DBP) and heart rate (HR), at: Pre-dose baseline, and 15(±5) min and 360(±15) post-dose, at each Study Visit. | 360 minutes post dose
Post-dose 20(±5) min ECG recordings (Routine and QT, QTc analysis) at each Study Visit, compared to the Screening baseline recording. | 20 minutes post dose
Data for physical examinations, CBC, serum comprehensive metabolic panel, and urinalysis for all subjects, and urinary pregnancy test for women of child-bearing potential | Screening and end of study
Monitoring of adverse drug events (ADE) | Ongoing through End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Jim Shi, M.D., Ph.D., Study Chair — Amphastar Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Amphastar Site 0001, San Jose, California
  - Amphastar Site 0003, Stockton, California

REFERENCES:
- [Background] Pinnas JL, Schachtel BP, Chen TM, Roseberry HR, Thoden WR. Inhaled epinephrine and oral theophylline-ephedrine in the treatment of asthma. J Clin Pharmacol. 1991 Mar;31(3):243-7. doi: 10.1002/j.1552-4604.1991.tb04969.x. PMID 2019665
- [Background] Hendeles L, Marshik PL, Ahrens R, Kifle Y, Shuster J. Response to nonprescription epinephrine inhaler during nocturnal asthma. Ann Allergy Asthma Immunol. 2005 Dec;95(6):530-4. doi: 10.1016/S1081-1206(10)61014-9. PMID 16400891
- [Background] Warren JB, Doble N, Dalton N, Ewan PW. Systemic absorption of inhaled epinephrine. Clin Pharmacol Ther. 1986 Dec;40(6):673-8. doi: 10.1038/clpt.1986.243. PMID 3780129
- [Background] Cripps A, Riebe M, Schulze M, Woodhouse R. Pharmaceutical transition to non-CFC pressurized metered dose inhalers. Respir Med. 2000 Jun;94 Suppl B:S3-9. PMID 10919679
- [Background] Dickinson BD, Altman RD, Deitchman SD, Champion HC. Safety of over-the-counter inhalers for asthma: report of the council on scientific affairs. Chest. 2000 Aug;118(2):522-6. doi: 10.1378/chest.118.2.522. PMID 10936150
- [Background] Simons FE, Gu X, Johnston LM, Simons KJ. Can epinephrine inhalations be substituted for epinephrine injection in children at risk for systemic anaphylaxis? Pediatrics. 2000 Nov;106(5):1040-4. doi: 10.1542/peds.106.5.1040. PMID 11061773
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Crapo RO, Morris AH, Clayton PD, Nixon CR. Lung volumes in healthy nonsmoking adults. Bull Eur Physiopathol Respir. 1982 May-Jun;18(3):419-25. PMID 7074238
- [Background] Dauphinee B, Tashkin DP, et al: Placebo-controlled evaluation of the speed of onset of epinephrine metered-dose aerosol (Primatene Mist) in mild to moderate asthmatics. Am J Respir Crit Care Med, 149:A204, 1994
- [Background] Armstrong Pharmaceuticals: Package Insert of Epinephrine Inhalation Aerosol USP, a CFC-MDI, current as of 2008
- [Background] Westfall TC, Westfall DP: Adrenergic agonists and antagonists, in Brunton LL, Lazo JS, Parker KL (eds): Goodman & Gilman's Ther Pharmacological Basis of Therapeitucs, 11th Ed. P237-296, 1986
- [Background] Montreal Protocol on substances that deplete the ozone layer, Montreal, Spet 1987; Adjusted and/or amended in London 1990; Copenhagen 1992; Vienna 1995; Montreal 1997 and Beijing 1999.
- [Background] NHLBI/NAEPP (National Heart, Lund and Blood Institute; Natuinak /asthma Education and Prevention Program) Expert Panel Report 3 (2007): Guidelines for the diagnosis and management of asthma, Section 3, Component 1, Figure 3-4C:
- [Background] Wyeth Consumer Healthcare: 2005N-0374, Use of ozone-depleting substances: Essential-use determination of over-the-counter (OTC) epinephrine metered dose inhalers. Submitted to teh Nonprescription Drugs and Pulmonary-Allergy Drugs Advisory Committees. Dec 2005.
- [Background] Global Initiative for Asthma (GINA): Pocket guide for asthma management and prevention,
- [Derived] Kerwin EM, Tashkin DP, Murphy TR, Bensch GW, Marrs T, Luo MZ, Zhang JY. A Dose-Ranging Study of Epinephrine Hydrofluroalkane Metered-Dose Inhaler (Primatene(R) MIST) in Subjects with Intermittent or Mild-to-Moderate Persistent Asthma. J Aerosol Med Pulm Drug Deliv. 2020 Aug;33(4):186-193. doi: 10.1089/jamp.2019.1558. Epub 2020 Mar 6. PMID 32150492